CLINICAL TRIAL: NCT03766230
Title: Subclinical Sympathetic Response Related to Second-eye Pain in Cataract Surgery and Its Noninvasive Detection Index
Brief Title: Clinical Study on Second-eye Pain in Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: YFZX2018006
Record Dates: First submitted 2018-08-19; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Senile Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The aqueous humor will be obtained in the surgery and kept in centrifugal tube. The amount of inflammatory cytokines will be measured afterwards.

GROUPS / COHORTS (10):
- peribulbar anesthesia1: Time interval between two eyes' cataract surgery is or less than 14 days and using peribulbar anesthesia
- topical anesthesia1: Time interval between two eyes' cataract surgery is or less than 14 days and using topical anesthesia
- peribulbar anesthesia2: Time interval between two eyes' cataract surgery is from 15 to 21 days and using peribulbar anesthesia
- topical anesthesia2: Time interval between two eyes' cataract surgery is from 15 to 21 days and using topical anesthesia
- peribulbar anesthesia3: Time interval between two eyes' cataract surgery is from 22 to 28 days and using peribulbar anesthesia
- topical anesthesia3: Time interval between two eyes' cataract surgery is from 22 to 28 days and using topical anesthesia
- peribulbar anesthesia4: Time interval between two eyes' cataract surgery is from 29 to 60 days and using peribulbar anesthesia
- topical anesthesia4: Time interval between two eyes' cataract surgery is from 29 to 60 days and using topical anesthesia
- peribulbar anesthesia5: Time interval between two eyes' cataract surgery is from 61 to 90 days and using peribulbar anesthesia
- topical anesthesia5: Time interval between two eyes' cataract surgery is from 61 to 90 days and using topical anesthesia

SUMMARY:
The degree of perceived pain in the second-eye surgery of cataract patients is significantly higher than that in the first-eye surgery, which can lead to nervous tension during surgery and affect the surgical outcome and satisfaction. Study suggested that in addition to psychological factors, there might be subclinical sympathetic reactions leading to increased pain in the second-eyes, but the objective indicators and clinical relevance are not clear. Therefore, it is necessary to study the mechanism of second-eye pain in cataract surgery, and to provide a test index that can effectively predict the degree of intraoperative pain in patients, as an important reference for the development of a suitable time for second eye surgery.

This study is based on clinical case studies, recruiting patients with clinically diagnosed binocular age-related cataract and require binocular surgery, to compare the correlation of intraocular inflammatory factors in the second eye and patients' self-pain scores while both eyes' surgery are completed by the same doctor in the same operating room, and the correlation of the change of inflammatory factors and the time interval between the two eyes surgery, to analyze the second-eye subclinical sympathetic reaction changing with the time interval after the first cataract surgery from the molecular biological results. Using the latest international anterior segment vascularization optical coherence tomography(OCT) scan and optical microvascular imaging(OMAG) analysis technology to quantify iris blood flow, this study analyzes the iris blood flow density, vascular density and other indicators before and after cataract surgery, and carry out its correlation with the degree of intraocular subclinical sympathetic reaction, providing a rapid, non-invasive objective examination index of the second-eye subclinical sympathetic response.

DETAILED DESCRIPTION:
1. Coordination and Quality Control Team: The inspection and audit of this research project will be established mainly by hospital clinical research center staff and assisted by the Ophthalmology Reading Center team;
2. The project team member will accept training before the study begins while unified inspection methods and requirements is established in standard operating procedures.
3. The project team double enter the test data independently and establishes an electronic database.
4. The project team randomly selects the data and repeats the measurements to ensure the accuracy as internal audit regularly.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with binocular age-related cataract.
2. Both eyes require phacoemulsification and intraocular lens implantation.
3. binocular surgery was performed by the same physician in the same operating room, and the anesthesia and surgical procedures were consistent.
4. Patients can fully understand the research purpose, research content, accidents and benefits and risks of the clinical trial, and can make their own decisions on participating or not.

Exclusion Criteria:

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Binocular senile cataract patients with binocular phacoemulsification and intraocular lens implantation to be performed at the Department of Ophthalmology in Shanghai Eye Disease Prevention and Treatment Center or Shanghai General Hospital from August 2018 to August 2020.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Surgery Pain Severity Score | Within one hour after first eye surgery; within one hour after second eye surgery (performed up to 90 days after first eye surgery)
  visual analogue scale is used to assess the surgery pain. Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients. A VAS is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling, the position of the respondent's cross is generally assigned a score between 0 and 100.

SECONDARY OUTCOMES:
Change in Concentration of inflammatory factors in aqueous humor | aqueous humor is acquired at the beginning of the first eye surgery and the second eye surgery (performed up to 90 days after first eye surgery)
  the Concentrations of tumor necrosis factor-α,interleukin-1,interleukin-6,interleukin-8,monocyte chemotactic protein-1,interleukin2,macrophage inflammatory protein-1α,macrophage inflammatory protein-1,carbon tetrachloride ,chemokine ligand 9,Tissue inhibitor of matrix metalloproteinase 01,C-C motif chemokine 11 are measured using Luminex
Change in blood flow density of iris vascular | Within 24 hours before first eye surgery and Day 1, Week 1, Week 3, Month 1, Month 3 after first eye surgery, or within 24 hours before second-eye surgery (performed up to 90 days after first eye surgery)
  CIRRUS High Definition-OCT 5000(Carl Zeiss Meditec, Dublin, CA)
Change in vascular density of iris vascular | Within 24 hours before first eye surgery and Day 1, Week 1, Week 3, Month 1, Month 3 after first eye surgery, or within 24 hours before second-eye surgery (performed up to 90 days after first eye surgery)
  CIRRUS High Definition-OCT 5000(Carl Zeiss Meditec, Dublin, CA)

IPD SHARING:
Plan to Share IPD: Undecided